CLINICAL TRIAL: NCT05599412
Title: A Prospective, Single-arm, Open-label, Non-interventional, Multi-centre, Post Marketing Surveillance (PMS) Study of Lorviqua (Registered)
Brief Title: Post Marketing Surveillance(PMS) Study of Lorviqua in Korea
Status: Recruiting | Type: Observational
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: B7461034; NCT05599412 (Registry Identifier: ClinicalTrials.gov)
Record Dates: First submitted 2022-10-26; First posted 2022-10-31 (Actual); Last update posted 2025-03-12 (Actual); Status verified 2025-03

CONDITIONS: Metastatic ALK+ Non Small Cell Lung Cancer

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Korean patients with Metastatic ALK+ Non small cell lung cancer
  Interventions: Drug: Lorviqua

INTERVENTIONS:
Drug: Lorviqua — As provided in real world practice

SUMMARY:
The objective of this study is to monitor the usage of Lorviqua in real practice within label, including the adverse events associated with Lorviqua

ELIGIBILITY:
Inclusion Criteria:

Patients must meet all of the following inclusion criteria to be eligible for inclusion in the study:

1. Use in the treatment of adult patients with anaplastic lymphoma kinase (ALK)-positive metastatic non-small cell lung cancer (NSCLC)
2. Evidence of a personally signed and dated informed consent document indicating that the patient (or a legally acceptable representative) has been informed of all pertinent aspects of the study.

Exclusion Criteria:

Patients meeting any of the following criteria will not be included in the study:

1. Patients to whom Lorviqua® is contraindicated as per the local labeling. A. Hypersensitivity to Lorviqua® or to any of the excipients of this product B. Lorviqua® is contraindicated in patients taking concomitant use of strong CYP3A4/5 inducers C. This medicinal product contains lactose as an excipient. Patients with rare hereditary problems of galactose intolerance, total lactase deficiency, or glucose galactose malabsorption should not take this medicinal product.
2. Any patients (or a legally acceptable representative) who does not agree that Pfizer and companies working with Pfizer use his/her information

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Korean patient who has a disease for which Lorlatinib is indicated
Sampling Method: Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2023-05-22 (Actual); Primary Completion 2028-03-31 (Estimated); Study Completion 2028-03-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of the adverse events from baseline | Up to 2 years
  This is a prospective, observational, non-interventional, multi-center study in which subjects will be administered as part of routine practice at Korean health care centers by accredited physicians.

SECONDARY OUTCOMES:
Objective Response Rate (ORR) per Response Evaluation Criteria in Solid Tumors (RECIST 1.1) | Up to 2 years
  To assess the effectiveness of Lorviqua® in patients with ALK-positive metastatic NSCLC under routine clinical practice in Korea.
Partial Response (PR) | Up to 2 years
Stable Disease (SD) | Up to 2 years
Progressive Disease (PD) | Up to 2 years
Complete Response (CR) | Up to 2 Years

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=B7461034